CLINICAL TRIAL: NCT02719652
Title: Vessel Wall and Perfusion Imaging in Intracranial Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiuhai Guo (Other)
Responsible Party: Sponsor-Investigator, Xiuhai Guo, Director of Clinical Research, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: ICAD-001
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-03

CONDITIONS: Intracranial Atherosclerosis
Keywords: intracranial atherosclerotic disease（ICAD）; vulnerable plaque; high-resolution magnetic resonance imaging （HR-MRI）
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- symptomatic ICAD: symptomatic intracranial atherosclerosis diseases
- asymptomatic ICAD: asymptomatic intracranial atherosclerosis diseases

SUMMARY:
Intracranial atherosclerotic disease (ICAD) is an important cause of ischemic stroke. The occurrence of stroke caused by symptomatic ICAD is significantly different compared with asymptomatic ICAD (19% vs 3.5%), suggesting that plaque vulnerability may be responsible for the difference. Based on the previous high-resolution magnetic resonance vessel wall imaging (HR-MRI) results, the investigators hypothesis that the feature of intracranial plaque enhancement is an important imaging biomarker of plaque instability, which is closely related to stroke. The investigators will establish the ICAD cohort and use HR-MRI to investigate the composition, morphology and the enhancement pattern of symptomatic ICAD plaques. These findings will correlate with biochemical markers, and stroke recurrence, in order to explore:

1. plaque characteristics and the enhancement features between symptomatic ICAD and asymptomatic ICAD
2. the relationship between plaque enhancement and the composition of plaques;
3. relationship among enhancement features of symptomatic ICAD plaques, biomarkers with different clinical significance,
4. evolution of enhancement features of symptomatic ICAD plaques under intensive medical therapy.

The investigators aim to explore the correlation between vulnerable plaque stratification and clinical outcomes, to explore the value of vascular responses in the pathogenicity of ICAD vulnerable plaques, as well as to provide objective basis for the establishment of the evaluation criteria of intracranial atherosclerotic vulnerable plaques.

DETAILED DESCRIPTION:
Detailed description:

Title: Vessel wall and Perfusion Imaging in Intracranial Atherosclerosis

Design: This is an prospective study that will study the characteristics of intracranial atherosclerotic plaque and the enhancement features of symptomatic ICAD during a mean follow-up of 1 year in symptomatic or asymtomatic patients with moderate to severe stenosis of middle cerebral artery(MCA).

In the WASID trail,patients with at least 70% stenosis of a major intracranial artery had an increased risk of recurrent stroke. However,The degree of stenosis is no longer the single predictor of vulnerable atherosclerotic lesions. Vulnerable plaques are closely associated with stroke recurrence.With the development of neurologic imaging, HR-MRI has unique ability to provide information on plaque compositions, plaque burden and vulnerable features. Several recent investigations suggest that enhancement of intracranial plaque is associated with recurrent stroke. However, no corhort study has been performed.

This prospective, multicenter trail will be conducted in China. Based on the previous work,participants will be divided into two groups :symtomatic ICAD and asymtomatic ICAD. Neurological examination and clinical sera testing will be performed at baseline, 1 month, 3 months, 6 months, and 12 months.The stroke incidence rate of asymptomatic ICAD and stroke recurrence rate of symptomatic ICAD will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients who suffered TIA or non-severe ischemic stroke(NHISS ≤6) in one week with 50% to 90% stenosis of MCA.
* Asymptomatic patients with ≥50% MCA stenosis without history of cerebrovascular events or an ischemic event in a territory outside that supplied by the affected MCA.
* Degree of ≥50% stenosis must be conformed by MRA, CTA and/or TCD.
* Age: 18-80 years.
* mRS scale score of ≤2.
* Patients who agree with future follow-up visits.
* Patients who sign the informed consent.

Exclusion Criteria:

* Coexistent ipsilateral internal carotid stenosis（≥50%）on MRA, CTA and/or TCD. Non-atherosclerotic vasculopathy, such as dissection, vasculitis,or moyamoya disease.
* Evidence of cardioembolism, such as atrial fibrillation, mechanical prosthetic valve disease, sick sinus syndrome, dilated cardiomyopathy, left ventricular thrombus, or recent myocardial infarction, hemorrhage, watershed infarction, or other cerebral diseases, such as vascular malformation, neoplasms, and encephalopyosis.
* Patients who are unable to undergo HR-MRI owing to underlying medical conditions.
* Patients who are allergic to any of the study medications, including aspirin, clopidogrel,atorvastatin,or rosuvastatin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with significant MCA stenosis（≥50%）on TCD, MRA, and/or CTA together with one or more risk factors of atherosclerosis will be prospectively recruited. Symtomatic patients will be included if they had suffered from a recent transient ischemic attack or ischemic stroke(NHISS≤6) in the territory of the stenotic MCA. Asymptomatic patients will be included if they had no history of cerebrovascular events or a history of an ischemic event in a territory outside that the affected MCA.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Stroke recurrence | 1 year
  the number of symptomatic participants who suffer from stroke recurrence after enrollment in the territory of the stenotic MCA.

SECONDARY OUTCOMES:
Death | 1 year
  The number of participants who suffer from death after enrollment
Any stroke, severe transient ischemic attack (TIA) outside the territory of symptomatic MCA | at 7 days, 30 days,3 months，6 months, 12 months
  The number of participants who suffer from any stroke, severe transient ischemic attack (TIA) outside the territory of symptomatic MCA
Stroke of asymptomatic participants | 1 year
  The number of asymptomatic participants who suffer from stroke after enrollment in the territory of the stenotic MCA；

CONTACTS AND LOCATIONS:
Overall Officials: Guo Xiuhai, MD, Principal Investigator — Xuanwu Hospital, Capital Medical University, Beijing, China; Qi Yang, MD, Principal Investigator — Xuanwu Hospital, Capital Medical University, Beijing, China
Locations (1):
- Department of Neurology, Xuanwu hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The date of individual participant will be recorded in case report form(CRF),which will be stored technically

REFERENCES:
- [Result] Mossa-Basha M, Hwang WD, De Havenon A, Hippe D, Balu N, Becker KJ, Tirschwell DT, Hatsukami T, Anzai Y, Yuan C. Multicontrast high-resolution vessel wall magnetic resonance imaging and its value in differentiating intracranial vasculopathic processes. Stroke. 2015 Jun;46(6):1567-73. doi: 10.1161/STROKEAHA.115.009037. Epub 2015 May 7. PMID 25953365
- [Result] Ahn SH, Lee J, Kim YJ, Kwon SU, Lee D, Jung SC, Kang DW, Kim JS. Isolated MCA disease in patients without significant atherosclerotic risk factors: a high-resolution magnetic resonance imaging study. Stroke. 2015 Mar;46(3):697-703. doi: 10.1161/STROKEAHA.114.008181. Epub 2015 Jan 27. PMID 25628303
- [Result] Ryoo S, Cha J, Kim SJ, Choi JW, Ki CS, Kim KH, Jeon P, Kim JS, Hong SC, Bang OY. High-resolution magnetic resonance wall imaging findings of Moyamoya disease. Stroke. 2014 Aug;45(8):2457-60. doi: 10.1161/STROKEAHA.114.004761. Epub 2014 Jun 19. PMID 24947295
- [Result] Holmstedt CA, Turan TN, Chimowitz MI. Atherosclerotic intracranial arterial stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2013 Nov;12(11):1106-14. doi: 10.1016/S1474-4422(13)70195-9. PMID 24135208
- [Result] Vakil P, Vranic J, Hurley MC, Bernstein RA, Korutz AW, Habib A, Shaibani A, Dehkordi FH, Carroll TJ, Ansari SA. T1 gadolinium enhancement of intracranial atherosclerotic plaques associated with symptomatic ischemic presentations. AJNR Am J Neuroradiol. 2013 Dec;34(12):2252-8. doi: 10.3174/ajnr.A3606. Epub 2013 Jul 4. PMID 23828109